CLINICAL TRIAL: NCT06682871
Title: The Effect Of Post-Birth Analgesia Interventions Performed To Purposed Of Elective Cesarean Delivery With Spinal Anesthesia In Our Hospital On The Initiating Of Breastfeeding And Exclusive Breastfeeding.
Brief Title: Breastfeeding Evaluation of Puerperal Women Who Had Cesarean Delivery in Our Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, RAMAZAN KEÇECİ, NEONATOLOGIST, MD, PRINCIPAL INVESTIGATOR, Konya City Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024/4806
Record Dates: First submitted 2024-10-21; First posted 2024-11-12 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Breast Feeding; Analgesia
Keywords: Post-cesarean analgesia; Breastfeeding; latch score; visuel pain score
MeSH Terms: conditions — Breast Feeding; Agnosia | interventions — Analgesia

STUDY DESIGN:
Intervention Model Description: D. Protocol After eligibility is confirmed, patients will receive complete information about the study both verbally and in writing. Informed consent will be obtained from the patients prior to randomization and study-specific procedures.
  Randomization will be based on computer-generated codes and use random-sized blocks. Allocations will be concealed until the morning of surgery where they will be provided by a web-based system.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be based on computer-generated codes and use random-sized blocks. Allocations will be concealed until the morning of surgery where they will be provided by a web-based system
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm T: Transversus Abdominis Plane (TAP) blocks with bupivacaine (Active Comparator): Infants of mothers who received 4-Quadrant TAP block after inactive elective spinal cesarean section (25 patients)
  Interventions: Procedure: Analgesia
- Arm E : Epidural Analgesia with bupivacaine (Active Comparator): Infants of mothers who received Epidural analgesia after inactive elective spinal cesarean section (25 patients)
  Interventions: Procedure: Analgesia
- Arm M: Iv Multimodal Analgesia with paracetamol or tramadol (Active Comparator): Infants of mothers who received Multimodal intravenous analgesia after inactive elective spinal cesarean section (25 patients)
  Interventions: Procedure: Analgesia

INTERVENTIONS:
Procedure: Analgesia — Postoperatively, patients will be given analgesia

SUMMARY:
İntroduction The World Health Organisation (WHO) and United Nations Children's Fund (UNICEF) recommends that infants are exclusively breastfed for a minimum of 6 months, with continued breastfeeding recommended until child age of 2 years or over to optimize growth, development, and health. Breast milk shows significant benefits for the physical and mental health of mothers and infants, including the promotion of maternal and infant bonding, the reduction of neonatal mortality, the reduction of maternal postoperative complications, and the development of newborns. Breastfeeding has been associated with improved maternal/infant bonding and increased child intelligence.

It is also clear that medical interventions during labor and birth, including a caesarean section, impact on women's infant feeding decisions and are a cause for concern given increasing global caesarean birth rates, with woman who have a planned caesarean birth reported as less likely to intend to breastfeed than women who did not have a planned caesarean birth or had a vaginal birth. Infrequent feeding and women's limited mobility in the early days following surgery may impede efforts to provide basic infant care. High levels of postoperative pain, particularly in the first 24 hrs, were also found to have a negative impact on women's breastfeeding experiences. Cesarean delivery is linked with lower rates of early breastfeeding initiation.

Pain management after casarean delivery remains challenging. The best-accepted traditional analgesic approach is continuous epidural analgesia. However, epidural analgesia is rapidly being replaced by transversus abdominis plane (TAP) blocks. TAP infiltration is an alternative to epidural blocks for providing postoperative analgesia to the anterior abdominal wall. TAP infiltrations are relatively easy to perform, generally safe, and can be performed in patients who are anti-coagulated. TAP infiltration can be performed as a single injection, or a catheter can be inserted for continuous local anesthetic infusion.

DETAILED DESCRIPTION:
İntroduction The World Health Organisation (WHO) and United Nations Children's Fund (UNICEF) recommends that infants are exclusively breastfed for a minimum of 6 months, with continued breastfeeding recommended until child age of 2 years or over to optimize growth, development, and health. Breast milk shows significant benefits for the physical and mental health of mothers and infants, including the promotion of maternal and infant bonding, the reduction of neonatal mortality, the reduction of maternal postoperative complications, and the development of newborns. Breastfeeding has been associated with improved maternal/infant bonding and increased child intelligence. In addition breastfeeding has many benefits for infant, mother and later child health.

The World Health Organization (WHO) and the United Nations Children's Fund (UNICEF) recommend initiation of breastfeeding within the first hour of birth, referred to as "early initiation of breastfeeding." Early initiation of breastfeeding is critical to newborn survival and to establish breastfeeding practice over the long term. When breastfeeding is delayed after birth, the consequences can be life-threatening and the longer newborns are left waiting, the greater the risk.

It is also clear that medical interventions during labor and birth, including a caesarean section, impact on women's infant feeding decisions and are a cause for concern given increasing global caesarean birth rates, with woman who have a planned caesarean birth reported as less likely to intend to breastfeed than women who did not have a planned caesarean birth or had a vaginal birth. Infrequent feeding and women's limited mobility in the early days following surgery may impede efforts to provide basic infant care. High levels of postoperative pain, particularly in the first 24 hrs, were also found to have a negative impact on women's breastfeeding experiences. Cesarean delivery is linked with lower rates of early breastfeeding initiation.

Pain management after casarean delivery remains challenging. The best-accepted traditional analgesic approach is continuous epidural analgesia. However, epidural analgesia is rapidly being replaced by transversus abdominis plane (TAP) blocks. TAP infiltration is an alternative to epidural blocks for providing postoperative analgesia to the anterior abdominal wall. TAP infiltrations are relatively easy to perform, generally safe, and can be performed in patients who are anti-coagulated. TAP infiltration can be performed as a single injection, or a catheter can be inserted for continuous local anesthetic infusion.

We therefore proposed to compare impact of TAP block, epidural analgesia and iv multimodal analgesia after spinal analgesia on maternal comfort in patients with elective caesarean section. We will evaluate the following specific aims, all of which will be assessed over 72 hours, or the duration of hospitalization if shorter:

Primary Aim: To compare the effect of pain management after cesarean on the rates of initiation of breastfeeding in the first hour after birth and exclusive breast milk in the first 72 hours in elective cesarean deliveries with spinal anesthesia.

Secondary Aim 1: To compare the effect of pain management after cesarean on the rates of the confidence and comfort of breastfeeding mothers after elective cesarean deliveries with spinal anesthesia.

Hypothesis. Four quadrant TAP blocks performed after elective inert cesarean section increase the rate of breastfeeding in the first 1 hour and the rate of exclusive breastfeeding in the first 72 hours.

3. Method and Study Design A. Study Overview A randomized double-blind trial is designed comparing TAP blocks , epidural analgesia and ıv multimodal analgesia and placebo in patients having elective inert cesarean deviveries with spinal anesthesia. The study will be performed at Konya City Hospital with IRB approval and written consent from patients.

B. Setting and Population

Inclusion criteria:

* Written informed consent;
* 18-45 years old;
* ASA Physical Status 1-3;
* Scheduled for elective cesarien delivery;
* Anticipated hospitalization of at least three nights;
* Expected requirement for parenteral opioids for at least 72 hours for postoperative pain;
* Able to use IV PCA systems.

Exclusion criteria:

* Hepatic disease, e.g. twice the normal levels of liver enzymes;
* Kidney disease, e.g. twice the normal level of serum creatinine;
* Bupivacaine sensitivity or known allergy;
* Anticoagulants considered to be a contraindication for TAP blocks;
* Surgeries with high port sites;

C. Withdrawal Criteria Patients will be free to withdraw from study at any time. Patients will also be removed from study at any time for adverse events, or deemed necessary for patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent;
* 18-45 years old;
* ASA Physical Status 1-3;
* Scheduled for elective cesarien delivery;
* Anticipated hospitalization of at least three nights;
* Expected requirement for parenteral opioids for at least 72 hours for postoperative pain;
* Able to use IV PCA systems.

Exclusion Criteria:

* Hepatic disease, e.g. twice the normal levels of liver enzymes;
* Kidney disease, e.g. twice the normal level of serum creatinine;
* Bupivacaine sensitivity or known allergy;
* Anticoagulants considered to be a contraindication for TAP blocks;
* Surgeries with high port sites

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
To compare the effect of pain management after cesarean on the rates of initiation of breastfeeding | 1 year
  Four quadrant TAP blocks performed after elective inert cesarean section increase the rate of breastfeeding in the first 1 hour and the rate of exclusive breastfeeding in the first 72 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Keçeci, Specialist, Principal Investigator — Konya City Hospital
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The protocol can be shared once the study is completed
Supporting Information: Study Protocol
Time Frame: 1 year
Access Criteria: No Criteria
URL: https://pubmed.ncbi.nlm.nih.gov/

REFERENCES:
- [Result] MacGregor E, Hughes M. Breastfeeding experiences of mothers from disadvantaged groups: a review. Community Pract. 2010 Jul;83(7):30-3. PMID 20701189
- See also: PUBMED — https://pubmed.ncbi.nlm.nih.gov/